CLINICAL TRIAL: NCT02536053
Title: Functional Outcomes and Health Related Quality of Life in Lower Extremity Soft Tissue Sarcoma Patients After Limb Salvage: A Prospective Study
Brief Title: Outcomes in Lower Extremity Soft Tissue Sarcoma Patients After Limb Salvage
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, MD, Helsinki University Central Hospital
Other Study IDs: 324/13/03/02/2014/2
Record Dates: First submitted 2015-08-18; First posted 2015-08-31 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Limb Salvage
Keywords: [E04.100.814.603]
MeSH Terms: interventions — Limb Salvage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Limb salvage

SUMMARY:
This study aims to:

1. validate the Finnish version of the Musculoskeletal Tumor Society scale and the Toronto Extremity Salvage Score lower extremity sections and to
2. assess the functional ability and health-related quality of life (HRQoL) of lower extremity sarcoma patients who have undergone limb salvage surgery.

DETAILED DESCRIPTION:
The first purpose of this study is to validate the Finnish version of the Musculoskeletal Tumor Society scale and the Toronto Extremity Salvage Score upper extremity sections. The second purpose is to chart the functional capabilities and health-related quality of life (HRQoL) of upper extremity sarcoma patients who have undergone limb salvage surgery with local or free flaps.

Patient hospital records are retrospectively reviewed to chart the demographic and clinical data.

The recruitment of patient takes place at the outpatient clinic of Department of Oncology, Helsinki University Hospital. The study includes a cross-sectional assessment at one year follow-up with five validated questionnaires. A follow-up is conducted three years after surgery in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity soft tissue sarcoma locating in between hip/gluteus to foot
* No metastasis at the time of diagnosis
* Undergone limb salvage surgery
* A minimum of 1 year follow-up
* Written consent
* Age > 18

Exclusion Criteria:

* Age <18
* No limb-salvage surgery due to sarcoma

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lower extremity sarcoma patient who underwent limb-salvage surgery
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-12; Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Validity of the lower-limb Musculoskeletal Tumor Society score and the Toronto Extremity Salvage Score | two to five years
  The validity is studied
Reliability of the lower-limb Musculoskeletal Tumor Society score and the Toronto Extremity Salvage Score | two to five years
  The test-retest reliability is studied
Health-related quality of life after limb salvage | two to five years
  Assessment of health-related quality of life
Assessment of the functional ability after limb salvage | two to five years
  Assessment of functional ability

SECONDARY OUTCOMES:
Quality of Life Questionnaire-Core 30 | two to five years
  Health-related quality of life assessment
The 15-dimensions health-related quality of life instrument | two to five years
  Health-related quality of life assessment
The Musculoskeletal Tumor Society score lower extremity section | two to five years
  Functional assessment of the reconstructed limb
The Toronto Extremity Salvage Score lower extremity section | two to five years
  Functional assessment of the reconstructed limb

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD, PhD, Study Director — Helsinki University Hospital and University of Helsinki; Carl Blomqvist, MD, PhD, Study Director — Helsinki University Hospital and University of Helsinki
Locations (1):
- Cancer center, Helsinki University Hospital and University of Helsinki, Helsinki, Helsinki and Uusimaa, Finland